CLINICAL TRIAL: NCT03913065
Title: Head Computed Tomography for Predicting Neurological Outcome After Cardiac Arrest- a TTM-2 Substudy
Brief Title: Head Computed Tomography for Predicting Neurological Outcome After Cardiac Arrest
Status: Completed | Type: Observational
Sponsor: Lund University (Other)
Collaborators: Region Skane (Other); Charite University, Berlin, Germany (Other); Halmstad County Hospital (Other); Sahlgrenska University Hospital (Other); Karlstad Central Hospital (Other); Medical University Innsbruck (Other); University Hospital of Wales (Other); Hopital Lariboisière (Other); Nantes University Hospital (Other); University Hospital, Linkoeping (Other)
Responsible Party: Sponsor
Other Study IDs: TTM-2 CT-substudy
Record Dates: First submitted 2019-04-05; First posted 2019-04-12 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Heart Arrest, Out-Of-Hospital; Computed Tomography; Unconsciousness; Neurologic Deficits
Keywords: Cardiac arrest; Hypothermia; Neurological function; Cardiovascular disease; Cerebral oedema; Cerebral edema; Cerebral ischaemia; Cerebral ischemia; Gray-white-matter differentiation; Grey-white-matter differentiation; ROI; Regions of interest; CT; GWR; Neurological prognostication
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Unconsciousness; Neurologic Manifestations; Heart Arrest; Hypothermia; Cardiovascular Diseases; Brain Edema; Cerebral Infarction; Brain Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: None Retained — Serum samples collected in the main trial TTM-2 (ClinicalTrials.gov Identifier: NCT02908308)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Included patients: Cardiac arrest patients from sites participating in the TTM-2 CT-substudy still unconscious 48 hours after cardiac arrest are routinely examined with head computed tomography as soon as possible after inclusion.
  Interventions: Diagnostic Test: CT

INTERVENTIONS:
Diagnostic Test: CT — Head computed tomography on patients still unconscious 48 hours after cardiac arrest.Visual evaluation of generalized oedema ("eye-balling"). Manual and automated measurement of the differentiation of gray and white matter (GWR) using circular regions of interest (ROI).

SUMMARY:
The European Resuscitation Council (ERC) and the European Society of Intensive Care Medicine (ESICM) joint guidelines for post-resuscitation care recommend a multimodal approach to prognostication of neurological outcome.

However, head computed tomography (CT) which is commonly used for predicting long-term neurological outcome after cardiac arrest has not yet been examined prospectively in a clinical trial.

The primary purpose of the TTM-2 CT-substudy is to prospectively investigate and compare various methods of diagnosing generalized oedema on CT after cardiac arrest and it´s ability to predict long-term neurological outcome.

DETAILED DESCRIPTION:
This study is a sub-study to the international multicenter Targeted Hypothermia Versus Targeted Normothermia After Out-of-hospital Cardiac Arrest (TTM-2) Trial (ClinicalTrials.gov Identifier: NCT02908308).

All patients from participating centers still unconscious 48 hours after cardiac arrest will be routinely examined with CT. All other inclusion and exclusion criteria as well as treatment, neurological prognostication, withdrawal of life-sustaining therapy or follow-up will be handled according to TTM-2- protocol. Ethical approval for the main trial and this sub-study have been obtained from the Swedish Ethical Review Authority at Lund University (2015/228 and 2017/36). Both a patients´ next of kind or conscious patients have the opportunity to withdraw patients from the trial.

Pseudonymized original CT images will be uploaded to a two-way secured digital platform from Lund University (LUSEC). Two study radiologists blinded from clinical data will perform analyses according to protocol. Various methods of diagnosing generalized oedema will be investigated including eye-balling (oedema "yes"/"no"), as well as manual and automated measurements of the differentiation between the grey and white matter (GWR) by placing circular regions of interest (ROI). Primary outcome is the neurological outcome at 6 months after cardiac arrest using the modified Rankin Scale (mRS).

Secondary outcomes include neurocognitive outcomes such as the Glasgow Outcome Score-Extended version (GOS-E), Symbol-Digit-Modalities-Test (SDMT) and the Montreal Cognitive Assessment Score (MoCA).

The results of the radiological evaluations will also be correlated with other markers of neuronal injury such as biomarkers, clinical neurological information or neurophysiological examinations.

Additional analyses include evaluation of all available CT images of participating patients to investigate if there is any progression or regression of cerebral oedema.

ELIGIBILITY:
Inclusion Criteria:

* Out-of-hospital cardiac arrest
* Presumed cardiac cause of cardiac arrest
* Unconscious with a FOUR-score <M4 (not obeying verbal commands)
* Stable return of spontaneous circulation (20 min)
* Eligible for intensive care treatment without restrictions
* Inclusion within 180 minutes of ROSC
* Patient from participating centers, where head CT is routinely performed on all patients still unconscious 48 hours after cardiac arrest

Exclusion Criteria:

* Unwitnessed cardiac arrest with an initial rhythm of asystole
* Temperature on admission <30°C.
* Obvious or suspected pregnancy
* Intracranial bleeding
* On ECMO prior to ROSC
* Severe chronic obstructive pulmonary disorder (COPD) with long-term home oxygen therapy
* Patients from centers not participating in the TTM-2 CT-substudy
* Patients from participating centers not examined with head CT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with Out-of hospital cardiac arrest included in the TTM-2 trial and randomized to either targeted temperature management at 33°C or early treatment of fever.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2017-11-18 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-12 (Actual)

PRIMARY OUTCOMES:
Poor functional outcome | 180 days
  Assessed using the modified Rankin Scale (mRS), with a score of 4-6 being a poor outcome.

SECONDARY OUTCOMES:
Exploratory: Neurocognitive outcome | 180 days
  Montreal Cognitive Assessment Scale (MoCA), ranges from 0-30, a score above 26 is considered normal.
Exploratory: Neurocognitive outcome | 180 days
  Symbol Digit Modalities Test (SDMT)
Exploratory: Functional outcome | 180 days
  Glasgow Outcome Scale-Extended version (GOS-E)

CONTACTS AND LOCATIONS:
Overall Officials: Marion Moseby-Knappe, MD, Principal Investigator — Lund University and Skane University Hospitals Sweden; Tobias Cronberg, MD, PhD, Principal Investigator — Lund University and Skane University Hospitals Sweden
Locations (1):
- Marion Moseby-Knappe, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Moseby-Knappe M, Pellis T, Dragancea I, Friberg H, Nielsen N, Horn J, Kuiper M, Roncarati A, Siemund R, Unden J, Cronberg T; TTM-trial investigators. Head computed tomography for prognostication of poor outcome in comatose patients after cardiac arrest and targeted temperature management. Resuscitation. 2017 Oct;119:89-94. doi: 10.1016/j.resuscitation.2017.06.027. Epub 2017 Jul 4. PMID 28687281
- [Derived] Lang M, Kenda M, Scheel M, Martola J, Wheeler M, Owen S, Johnsson M, Annborn M, Dankiewicz J, Deye N, During J, Halliday T, Jakobsen JC, Lascarrou JB, Levin H, Lilja G, Lybeck A, McGuigan PJ, Rylander C, Sem V, Thomas M, Ullen S, Unden J, Wise MP, Cronberg T, Wasselius J, Nielsen N, Leithner C, Moseby-Knappe M. Radiological signs of hypoxic-ischaemic encephalopathy on head computed tomography for prediction of poor functional outcome after cardiac arrest - a prospective observational cohort study. Resuscitation. 2025 Sep;214:110675. doi: 10.1016/j.resuscitation.2025.110675. Epub 2025 Jun 9. PMID 40499676
- [Derived] Lang M, Leithner C, Scheel M, Kenda M, Cronberg T, During J, Rylander C, Annborn M, Dankiewicz J, Deye N, Halliday T, Lascarrou JB, Matthew T, McGuigan P, Morgan M, Thomas M, Ullen S, Unden J, Nielsen N, Moseby-Knappe M. Prognostic accuracy of head computed tomography for prediction of functional outcome after out-of-hospital cardiac arrest: Rationale and design of the prospective TTM2-CT-substudy. Resusc Plus. 2022 Oct 12;12:100316. doi: 10.1016/j.resplu.2022.100316. eCollection 2022 Dec. PMID 36267356
- See also: Website of the TTM2 trial — http://ttm2trial.org